CLINICAL TRIAL: NCT05349266
Title: Assessment of Safety and Efficacy of ThisCART19A in Adult Patients With B Cells Non-Hodgkin's Lymphoma(B-NHL) After Failure of Autologous CAR-T Therapy
Brief Title: Assessment of Safety and Efficacy of ThisCART19A in Adult Patients With B-NHL After Failure of Autologous Chimeric Antigen Receptor T- Cell(CAR-T) Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, President/Proffessor, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT400-003
Record Dates: First submitted 2022-04-08; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ThisCART19A 2×10^6 cells/kg for dose level 1 (Experimental): Patients will receive 2×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A
- ThisCART19A 3×10^6 cells/kg as dose level 2 (Experimental): Patients will receive 3×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A
- Patients will receive 4×10^6 cells/kg as dose level 3 (Experimental): Patients will receive 4×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A

INTERVENTIONS:
Biological: ThisCART19A — each patient will receive a dose level per body weight(kg) for only once.

SUMMARY:
This is a phase I, single center study to assess the efficacy and safety of ThisCART19A in adult with Non-Hodgkins Lymphoma in China.

ELIGIBILITY:
Inclusion Criteria:

* Cellular or histopathological diagnosis of B-cell non-Hodgkin's lymphoma (B-NHL) includes: diffuse Large B-cell lymphoma (DLBCL), follicular lymphoma to DLBCL (tFL), follicular lymphatic (FL), Mantle cell lymphoma (MCL), primary Mediastinal Large B-cell lymphoma (PMBCL), etc.
* Failing to autologous CAR-T therapy.
* At least one available lesion to be assessed.
* Good organ function during screening.
* Should be confirmed Cluster of differentiation(CD)19 positive by biopsy for the patient who received target CD19 therapy before.

Exclusion Criteria:

* Allergic to preconditioning measures.
* Patients with other malignancies other than B-cell malignancies within 5 years prior to screening. Patients with cured skin squamous carcinoma, basal carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be recruited.
* Uncontrollable bacterial, fungal and viral infection during screening.
* Patients had pulmonary embolism within 3 months prior to enrollment.
* Had intolerant severe cardiovascular and cerebrovascular diseases and hereditary diseases prior to enrollment.
* Imaging confirmed the presence of central nervous system involvement (both primary and secondary) and obvious symptoms at the time of screening.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) or Human immunodeficiency virus (HIV) or Syphilis infection. HBV-DNA < 2000 IU/mL can be enrolled, but should admitted to use anti-virus drugs such as entecavir, tenofovir, etc, and supervisory the relative indication during the treatment.
* Had big lesion(single lesion diameter ≥10 cm).
* Bone marrow involvement≥5%.
* Receive allogeneic hematopoietic stem cell transplantation less than 100 days.
* Combined systemic steroid use (e.g., prednisone ≥20mg) within 3 days prior to screening. Or systemic diseases that require long-term use of immunization Inhibitor.
* Vaccinated with influenza vaccine within 2 weeks prior to lymphodepleting chemotherapy (Severe Acute Respiratory Syndrome-Corona virus disease 19 can be included, inactivated, live/non-live adjuvant vaccinations allowed to be included) .
* Patients who are receiving Graft versus host disease Hepatitis(GvHD) treatment; Patients without GvHD and who had stopped immunosuppressive drugs for at least 1 month were eligible for inclusion.
* Women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after cell infusion. Male subjects who plan pregnancy within 1 year after infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) observation in patient with NHL during dose escalation stage | 28 days
  DLT is defined as the incidence of severe adverse events related to ThisCART19A more than 33% in each dose level.
Objective Response Rate in patient with NHL during dose expansion stage | 12 months
  the incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as best response to treatment

SECONDARY OUTCOMES:
Objective Response Rate during dose escalation stage and expansion stage | 12 months
  the incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as best response to treatment
Duration of response(DOR) during dose escalation stage and expansion stage | 12 months
  The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR)
OS(overall survival) during dose escalation stage and expansion stage | 12 months
  Overall survival (OS) is defined as the time from the date of lymphodepletion until death from any cause.
Time to remission(TTR) during dose escalation stage and expansion stage | 12 months
  Time to remission(TTR) is defined as the time from the date of ThisCART19A infusion until the date of first remission.
Analysis the change characteristics of CART cell number and copy number during dose escalation and expansion stages | 6 months
  Track CAR T cells expansion in patients after infusion
Analysis the change characteristics of cytokines and immune effect cells number during dose escalation and expansion stages | 3 months
  Analysis the effect cells and cytokines in patient after infusion
Analysis the severity and Incidence of Adverse Events in each dose level during dose expansion stage | 3 months
  Including more than or equal to grade 3 adverse events graded according to the NCI CTCAE v5.0, or the adverse events with special attention
Analysis the immunogenicity(anti-therapeutic antibody and neutralizing antibody) of CAR-T cells after infusion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, Doctor, Principal Investigator — First hospital affiliated Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China